CLINICAL TRIAL: NCT05962021
Title: Neoadjuvant Toripalimab Plus Chemotherapy for Resectable Stage II-IIIB Non-squamous Non-small Cell Lung Cancer With EGFR Mutation: a Multicentre, Multi-cohort, Exploratory Study.
Brief Title: Neoadjuvant Toripalimab for Non-squamous NSCLC With EGFR Mutation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Principal Investigator, Yang Fan, MD, Professor of Thoracic Surgery, Peking University People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ISS-CO413
Record Dates: First submitted 2023-07-10; First posted 2023-07-27 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Non Squamous Non Small Cell Lung Cancer; EGFR Positive Non-small Cell Lung Cancer
Keywords: Non squamous non small cell lung cancer; EGFR Mutation; Neoadjuvant immuno-chemotherapy; Predictive and prognostic biomarker
MeSH Terms: interventions — toripalimab; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Patients were divided into the 19del and L858R groups according to their EGFR mutation status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 19DEL cohort (Experimental): Patients who participated in the trial with EGFR 19DEL mutation will be included in this arm.
  Interventions: Drug: Toripalimab plus Chemotherapy
- L858R cohort (Experimental): Patients who participated in the trial with EGFR L858R mutation will be included in this arm
  Interventions: Drug: Toripalimab plus Chemotherapy

INTERVENTIONS:
Drug: Toripalimab plus Chemotherapy — Therapy was administered on a 21-day regimen for 3 cycles, with Toripalimab (240mg, d1), carboplatin (AUC=5, d1) + pemetrexed (500 mg/m2, d1) for patients with lung adenocarcinoma and carboplatin (AUC=5, d1) + albumin-bound paclitaxel (260 mg/m2, d1) for patients with other subtypes.

SUMMARY:
This study was designed to investigate the efficacy and safety of neoadjuvant Toripalimab (anti-PD1) plus chemotherapy for patients with resectable II-IIIB non-squamous NSCLC harboring EGFR mutation, and to explore the potential predictive and prognostic biomarkers, aiming to provide more abundant evidences for the preoperative treatment decision of non-squamous NSCLC patients.

DETAILED DESCRIPTION:
Previous studies have confirmed the efficacy of neoadjuvant immunotherapy in NSCLC patients without driver gene mutation, while its efficacy in driver gene mutated patients is still controversial. This study was designed to investigate the efficacy and safety of neoadjuvant Toripalimab (anti-PD1) plus chemotherapy for patients with resectable II-IIIB non-squamous NSCLC harboring EGFR mutation, and to explore the potential predictive and prognostic biomarkers, aiming to provide more abundant evidences for the preoperative treatment decision of non-squamous NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed informed consent by the patient or legally acceptable representative;
2. Previously untreated, histologically confirmed resectable stage II-IIIA, IIIB(N2) (AJCC staging 8th edition) non-squamous non-small cell lung cancer;
3. Adequate tissue samples for PD-L1 immunohistochemical testing and gene mutations test by RT-pCR or NGS, or consent for blood RT-PCR or NGS if tissue samples are insufficient;
4. Harboring EGFR mutation (19del or L858R);
5. Aged 18-70 years, regardless of gender;
6. Eastern Cooperative Group (ECOG) Performance Status 0-1;
7. Acceptable cardiac function with a left ventricular ejection fraction >50%;
8. Acceptable respiratory function (FEV1>1.5L, DLCO>50%) and ability to tolerate radical lung cancer surgery;
9. Acceptable bone marrow haematopoiesis with leucocytes ≥ 4 x 10^9/L, neutrophils ≥ 1.5 x 10^9/L, haemoglobin ≥ 10g/dL and platelets ≥ 100 x 10^9/L;
10. Acceptable renal function with a glomerular filtration rate ≥ 60 mL/min;
11. Acceptable liver function with total bilirubin ≤ 1.5 x ULN, AST ≤ 3 x ULN, and ALT ≤ 3 x ULN;
12. Presence of measurable lesions as defined by RECIST 1.1 criteria;
13. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 3 days prior to the start of study treatment, and agree to use effective contraception for the duration of study drug use and for 120 days after the last dose. Women of childbearing potential were defined as sexually mature females who 1) had not undergone hysterectomy or bilateral oophorectomy and 2) had not experienced spontaneous menopause for 12 consecutive months (amenorrhea after cancer treatment did not preclude fertility) (menstruation had occurred at any time during the previous 12 consecutive months).

Exclusion Criteria:

1. Pathological histologically confirmed small cell lung cancer, squamous epithelial cell carcinoma and other pathological subtypes cannot be enrolled;
2. Patients with advanced or metastatic lung cancer, or unresectable lung cancer, or who have received previous systemic anti-tumour therapy such as immunotherapy, chemotherapy or targeted therapy cannot be enrolled;
3. Patients with a history of active autoimmune disease or autoimmune disease that is likely to recur cannot be enrolled;
4. Patients with active hepatitis B and C requiring relevant antiviral therapy need to have HBV-DNA <500 IU/ml and have been on anti-HBV treatment for at least 14 days prior to study entry and continue treatment during the treatment period; HCV RNA-positive patients should be excluded;
5. Patients who are allergic to chemotherapeutic agents such as carboplatin, paclitaxel, albumin paclitaxel, pemetrexed;
6. Patients with a history of allergy to monoclonal antibody drugs;
7. Patients who have previously received an allogeneic stem cell transplant or organ transplant；
8. Patients with mental illness or any other illness that makes it impossible to comply with treatment；
9. Patients who are unable or unwilling to sign the informed consent form；
10. Patients with comorbidities or other conditions that, in the opinion of the investigator, may affect compliance with the protocol or make them unsuitable for participation in this study.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | Within 1 week after surgery
  Pathologic complete response (pCR) rate is defined as the percentage of participants with no residual viable tumor in lung primary or lymph nodes as evaluated by blinded independent pathological review (BIPR).

SECONDARY OUTCOMES:
Major Pathologic Response (MPR) Rate | Within 1 week after surgery
  Major pathologic response (MPR) rate is defined as the percentage of participants with less than or equal to 10% of residual viable tumor in lung primary or lymph nodes as evaluated by blinded independent pathological review (BIPR). Viable tumors in situ carcinoma should not be included in MPR calculation.
Pathologic Complete Response (pCR) Rate in non-squamous NSCLC with different EGFR mutations status | Within 1 week after surgery
  Assessing pCR rates in the 19del and L858R groups separately.
Major Pathologic Response (MPR) Rate in non-squamous NSCLC with different EGFR mutations status | Within 1 week after surgery
  Assessing MRP rates in the 19del and L858R groups separately.
Pathologic Complete Response (pCR) Rate in non-squamous NSCLC with different PD-L1 expression levels | Within 1 week after surgery
  Assessing pCR rates in the PD-L1 TPS≥1% and PD-L1 TPS<1% groups separately.
Major Pathologic Response (MPR) Rate in non-squamous NSCLC with different PD-L1 expression levels | Within 1 week after surgery
  Assessing MRP rates in the PD-L1 TPS≥1% and PD-L1 TPS<1% groups separately.
Event-free Survival (EFS) | Up to 24 months after participation
  EFS is defined as the time from participation to any of the following events: progression of disease, recurrence disease, or death due to any cause. Progression/recurrence will be assessed either by biopsy assessed by local pathologist or by investigator-assessed imaging using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
The Safety and Tolerability | Up to 24 months after participation
  To assess the safety and tolerability of neoadjuvant immuno-chemotherapy in patients with resectable stage II-IIIB non-squamous non-small cell lung cancer harboring EGFR mutations, including as follows: number, frequency and proportion of patients with adverse events (AEs), serious adverse events (SAEs) and AEs of special interest (AESI) and on-study deaths.

CONTACTS AND LOCATIONS:
Overall Officials: Fan Yanf, M.D., Study Chair — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided